CLINICAL TRIAL: NCT02246712
Title: Influence of Uncontrolled Diabetes on the Kinetic Disposition, Metabolism and Pharmacokinetics-pharmacodynamics of Tramadol Enantiomers in Patients With Neuropathic Pain
Brief Title: Influence of Diabetes on Tramadol Pharmacokinetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Natalia Valadares de Moraes, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIABETRA
Record Dates: First submitted 2014-09-16; First posted 2014-09-23 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Neuropathic Pain; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: tramadol; pharmacokinetics; enantiomers; metabolism; diabetes
MeSH Terms: conditions — Neuralgia; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Blood Specimen Collection; Cytochrome P-450 CYP2D6; Cytochrome P-450 CYP3A; Cytochrome P-450 CYP2B6

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Active Comparator): Patients received a single oral dose of 100 mg racemic tramadol. Serial blood samples were collected up to 24 h after administration of the drug for pharmacokinetic study and for the analysis of noradrenaline in plasma. Pain was rated on a visual analog pain scale at the same time as blood sampling. CYP2D6 phenotype was evaluated using metoprolol as probe drug. CYP3A phenotype was evaluated using midazolam. Patients were genotyped for the single nucleotide polymorphism (SNP) 516G>T in CYP2B6 gene (CYP2B6 genotype).
  Interventions: Drug: Single oral dose of 100 mg racemic tramadol; Other: CYP2D6 phenotype; Other: CYP3A phenotype; Genetic: CYP2B6 genotype
- T2DM group (Experimental): Patients received a single oral dose of 100 mg racemic tramadol. Serial blood samples were collected up to 24 h after administration of the drug for pharmacokinetic study and for the analysis of noradrenaline in plasma. Pain was rated on a visual analog pain scale at the same time as blood sampling. CYP2D6 phenotype was evaluated using metoprolol as probe drug. CYP3A phenotype was evaluated using midazolam. Patients were genotyped for SNP 516G>T in CYP2B6 gene (CYP2B6 genotype).
  The diagnosis of type 2 DM was performed according to the American Diabetes Association (2010).
  Interventions: Drug: Single oral dose of 100 mg racemic tramadol; Other: CYP2D6 phenotype; Other: CYP3A phenotype; Genetic: CYP2B6 genotype
- T1DM group (Experimental): Patients received a single oral dose of 100 mg racemic tramadol. Serial blood samples were collected up to 24 h after administration of the drug for pharmacokinetic study and for the analysis of noradrenaline in plasma. Pain was rated on a visual analog pain scale at the same time as blood sampling. CYP2D6 phenotype was evaluated using metoprolol as probe drug. CYP3A phenotype was evaluated using midazolam. Patients were genotyped for SNP 516G>T in CYP2B6 gene (CYP2B6 genotype).
  The diagnosis of type 1 DM was performed according to the American Diabetes Association (2010).
  Interventions: Drug: Single oral dose of 100 mg racemic tramadol; Other: CYP2D6 phenotype; Other: CYP3A phenotype; Genetic: CYP2B6 genotype

INTERVENTIONS:
Drug: Single oral dose of 100 mg racemic tramadol — Serial blood samples were collected up to 24 h after drug administration; Pain was evaluated at the same time of blood sampling using visual analog scale
  Other Names: Tramadol treament; Blood sampling; Tramadol pharmacokinetics
Other: CYP2D6 phenotype — Patients were phenotyped using metoprolol (100 mg, single oral dose). Urine was collected up to 8 hours after metoprolol administration. Urinary concentrations of metoprolol and alfa-hydroxymetoprolol were determined by high performance liquid chromatography (HPLC), using fluorescence detector.
  CYP2D6 phenotyped was determined by alfa-hydroxymetoprolol/metoprolol urinary rato
  Other Names: CYP2D6 phenotyping; CYP2D6 in vivo activity
Other: CYP3A phenotype — A single oral dose of midazolam (15 mg) was administered to all patients. Serial blood samples were collected up to 6 hours after the administration of midazolam.
  The concentration of midazolam was determined in plasma in order to calculate midazolam clearance.
  The in vivo activity of CYP3A was evaluated by midazolam oral clearance.
  Other Names: CYP3A phenotyping; CYP3A in vivo activity
Genetic: CYP2B6 genotype — The single nucleotide polymorphism 516G>T in CYP2B6 gene was evaluated using polymerase chain reaction-restriction fragment length polymorphism (PCR-RFLP).
  Other Names: Genotype of SNP 516G>T in CYP2B6

SUMMARY:
This study aimed to investigate the influence of uncontrolled type 1 and type 2 diabetes mellitus (DM) on the kinetic disposition, metabolism and pharmacokinetics-pharmacodynamics of tramadol enantiomers in patients with neuropathic pain. Thus, nondiabetic patients (control group, n = 12), patients with type 1 DM (n = 9), and patients with type 2 DM (n = 9), all with neuropathic pain and phenotyped as extensive metabolizers of cytochrome P450 2D6 (CYP2D6) who were treated with a single oral dose of 100 mg racemic tramadol were investigated.

DETAILED DESCRIPTION:
Tramadol is a centrally acting analgesic that effectively relieves acute and chronic pain, including neuropathic pain in diabetic patients. The drug is available in clinical practice as a mixture of the (+)-tramadol and (-)-tramadol enantiomers. Tramadol is metabolized by CYP2D6 to O-desmethyltramadol (M1) and by cytochrome P450 3A (CYP3A4) and cytochrome P450 2B6 (CYP2B6) to N-desmethyltramadol (M2). Both tramadol enantiomers and (+)-M1 contribute to the analgesic activity of the drug: (+)-tramadol and the (+)-M1 metabolite act as -opioid receptor agonists; (+)-tramadol inhibits serotonin reuptake; and (-)-tramadol inhibits the reuptake of norepinephrine. This study investigated the influence of uncontrolled type 1 and type 2 diabetes mellitus (DM) on the kinetic disposition, metabolism and pharmacokinetics-pharmacodynamics of tramadol enantiomers in patients with neuropathic pain. Nondiabetic patients (control group, n = 12), patients with type 1 DM (n = 9), and patients with type 2 DM (n = 9), all with neuropathic pain and phenotyped as extensive metabolizers of CYP2D6, received a single oral dose of 100 mg racemic tramadol. Serial blood samples were collected up to 24 h after administration of the drug for pharmacokinetic study and for the analysis of noradrenaline in plasma. Pain was rated on a visual analog pain scale at the same time as blood sampling. The patients were evaluated for in vivo CYP3A activity using midazolam as a probe drug and genotyped for CYP2B6. Total and unbound plasma concentrations of the tramadol, M1 and M2 enantiomers were analyzed by liquid chromatography coupled to tandem mass spectrometry (LC-MS/MS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, both gender
* Patients with self-reported neuropathic pain (score >4 in a 0-10 visual analog scale)
* Patients with normal renal function (creatinine clearance >60 mL/min)

Exclusion Criteria:

* Patients with nociceptive somatic pain, visceral or autonomic associated during the study period;
* Patients with morbid obesity (BMI> 40), congestive heart failure, severe hypertension
* Patients who have had acute myocardial infarction or accident stroke less than 6 months of the period of investigation.
* Patients with chronic obstructive pulmonary disease
* Patients who were in use of analgesics, CYP2D6 inhibitors or CYP3A4 inducers or inhibitors were excluded.
* Pregnant and lactating patients were excluded.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Kinetic parameters (AUC, Cmax, Tmax, apparent total clearance, and apparent volume of distribution) of tramadol enantiomers were estimated. | Up to 24h after a single oral dose of tramadol (100 mg)

SECONDARY OUTCOMES:
Urinary concentration ratio (metoprolol/alfa-hydroxymetoprolol) as an in vivo measure of CYP2D6 activity | Up to 8h after metoprolol administration
  The CYP2D6 phenotype was determined by urinary concentration ratio metoprolol/alfa-hydroxymetoprolol
Clearance of midazolam as a measure of CYP3A in vivo activity | Up to 6h after midazolam administration
Pain scores on the visual analog scale | Up to 24h after a single oral dose of tramadol (100 mg)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia V de Moraes, PhD, Principal Investigator — Universidade Estadual Paulista Julio de Mesquita Filho
Locations (1):
- Universidade Estadual Paulista Julio de Mesquita Filho, Araraquara, São Paulo, Brazil

REFERENCES:
- [Result] de Moraes NV, Lauretti GR, Lanchote VL. Effects of type 1 and type 2 diabetes on the pharmacokinetics of tramadol enantiomers in patients with neuropathic pain phenotyped as cytochrome P450 2D6 extensive metabolizers. J Pharm Pharmacol. 2014 Sep;66(9):1222-30. doi: 10.1111/jphp.12255. Epub 2014 Apr 10. PMID 24717054
- [Result] de Moraes NV, Lauretti GR, Napolitano MN, Santos NR, Godoy AL, Lanchote VL. Enantioselective analysis of unbound tramadol, O-desmethyltramadol and N-desmethyltramadol in plasma by ultrafiltration and LC-MS/MS: application to clinical pharmacokinetics. J Chromatogr B Analyt Technol Biomed Life Sci. 2012 Jan 1;880(1):140-7. doi: 10.1016/j.jchromb.2011.11.033. Epub 2011 Nov 28. PMID 22173007